CLINICAL TRIAL: NCT01557816
Title: A Randomized, Double-Blind, Placebo-controlled Cross-over, Exploratory Trial of Naproxen to Evaluate Methods of Measuring Analgesic Effect in Osteoarthritis Pain of the Knee
Brief Title: Trial of Naproxen to Evaluate Various Methods of Measuring Analgesic Effect in Osteoarthritis Pain of the Knee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Analgesic Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALPMF-006-2010
Record Dates: First submitted 2012-02-21; First posted 2012-03-20 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-02

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; knee; Naproxen
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Naproxen; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naproxen (Active Comparator)
  Interventions: Drug: Naproxen; Drug: Placebo
- Placebo (Sham Comparator)
  Interventions: Drug: Naproxen; Drug: Placebo

INTERVENTIONS:
Drug: Naproxen — Naproxen for 7 days (3 days at 250 mg BID followed by 4 days at 500 mg BID) during either of the 2 treatment periods.
  Other Names: Aleve; Naprosyn
Drug: Placebo — Placebo for seven days given BID during either of the 2 treatment periods.
  Other Names: Sugar pill

SUMMARY:
This study aims to evaluate various methods of measuring pain relief in subjects who have chronic OA of the knee. After a 1 week of wash-out from existing therapy, subjects will be treated in a blinded fashion for 1 week with either naproxen (3 days at 250 mg twice a day followed by 4 days at 500 mg twice a day) or placebo. After the first week of treatment, subjects will have another week of wash-out followed by a second period of 1 week of the alternate treatment. Subjects will not be allowed to use oral non-steroidal anti-inflammatory drugs (NSAIDs) or other oral analgesics, or topical medications on their target knees during the study. Acetaminophen will be allowed as a rescue medication.

DETAILED DESCRIPTION:
This study aims to evaluate various methods of measuring pain relief in osteoarthritis (OA) of the knee. The duration of the study will be up to 5 weeks. Eligible subjects will have chronic OA of the knee. After meeting initial entry criteria and prior to randomization, there will be a 1 week wash-out from existing therapy. Subjects will then be treated in a blinded fashion for 1 week with either naproxen (3 days at 250 mg twice a day followed by 4 days at 500 mg twice a day) or placebo. After the first week of treatment, subjects will have a week of wash-out followed by a second period of 1 week of the alternate treatment. Subjects will not be allowed to use oral non-steroidal anti-inflammatory drugs (NSAIDs) or other oral analgesics, nor will they be allowed to use topical medications on their target knees during the study. Acetaminophen will be allowed as a rescue medication (as needed up to 2 g/day)but subjects will be told not to take acetaminophen at least 12 hours before study visits. Seventy (70) subjects will be randomized to ensure that 60 subjects complete both treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. Subject able to read, comprehend and sign written Informed Consent Form
2. Subject is 21 years old or older
3. If female, should be post-menopausal or has negative urine test
4. Subject has some degree of target joint pain for the last 3 months
5. Subject has to have 3 out of six:

   ( )Age > 50 ( )Morning stiffness < 30 minutes ( )Crepitus on active motion ( )Bony enlargement ( )No palpable warmth of synovium
6. Subject had an X-ray of the target knee showing evidence of OA within the past 3 years
7. Target joint does not contain any type of orthopedic and/or prosthetic device
8. Subject is ambulatory
9. Subject is in good general medical and psychological health, and is capable of completing study assessments and procedures.

Exclusion Criteria:

1. Subject had an x-ray of the target knee showing Kellgren-Lawrence grade 4
2. Subject has any pain syndrome that has the potential to confound the assessment of the target knee.
3. the subject has a documented history of an adverse reaction to NSAIDs or acetaminophen
4. Subject is pregnant or breast feeding
5. Subject has sitting systolic pressure > 180 mmHg or < 90mmHg, and/or a sitting diastolic pressure > 100 mmHg or < 50 mmHg at screening
6. Subject has mass body index (BMI) > 35 kg/m2.
7. Subject has a Hospital Anxiety and Depression Scale (HADS) score > 12 on either subscale or has an established history of major depressive disorder not controlled with medication
8. Subject has had an introduction of physiotherapy, acupuncture, or transcutaneous electrical nerve stimulation within 4 weeks before screening, or has no stable regimen of these modalities.
9. Subject has a clinically significant abnormalities in clinical chemistry, hematology, coagulation, or urinalysis.
10. Subject has a significant history or renal impairment
11. Subject has a positive urine drug screen for alcohol, illicit drugs or nonprescribed controlled substances
12. Subject has dermatological lesions of the target knee or ipsilateral elbow at the time of screening.
13. Subject is unable to discontinue all formulations of prior analgesics
14. Subject has received any investigational drug within 30 days prior to screening
15. Subject has a history of active peptic ulceration, gastrointestinal bleeding, esophageal, or gastric or duodenal ulcer within 3 months of screening
16. Subject has had a surgical intervention for any pain within 3 months of screening or plans for surgical intervention while in the study
17. Subject has a documented history of inflammatory arthritis, including rheumatoid arthritis.
18. Subject has received local corticosteroid injections, viscosupplementation, or arthrocentesis in the target joint within 3 months of screening
19. Subject has received oral or intramuscular corticosteroids within the past 30 days
20. Subject is involved in an ongoing or settled worker's compensation claim, disability, or litigation related to any pain problem
21. Subject had used opioids for pain more than 4 days in the week preceding screening
22. Subject has a history of alcohol or drug abuse/dependence/misuse within 2 years of screening
23. Subject has history of acute coronary syndrome, ischemic or hemorrhagic stroke, transient ischemic attack, or previous revascularization procedure to coronary or peripheral vasculature, or has a history of congestive heart failure within 5 years of screening
24. Subject has had axillary lymph nodes removed bilaterally
25. Subject has a disease-related or iatrogenic coagulopathy, or had been diagnosed with thrombocytopenia or a functional platelet disorder
26. The subject is currently on an aromatase inhibitor.
27. Subject has a history of any condition that, in the Investigator's opinion, precludes participation in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of naproxen vs. placebo | 5 weeks
  Efficacy of naproxen VS placebo will be analyzed by efficacy end-points of within-subject difference. Efficacy evaluations will include:
  * In-clinic pain intensity NRS (24-hour recall)
  * WOMAC: pain subscale, stiffness subscale, function subscale, and total scores
  * Daily actiwatch pain intensity
  * In-clinic pain intensity NRS for curent pain at rest and after exercise
  * Thermal pain matching at rest and after exercise
  * PGIC (Patient's Global Impression of Change)
  * Subject treatment reference
Safety | 5 weeks
  Safety of Naproxen VS Placebo
  Safety evaluations will include:
  * Adverse events (AEs)and serious AEs (SAEs)
  * Vital signs
  * Clinical Laboratories
  * Concomitant medications

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Wright, MD, Principal Investigator — Analgesic Solutions
Locations (1):
- Analgesic Solutions, Natick, Massachusetts, United States